CLINICAL TRIAL: NCT07350824
Title: Predictive Value of Minimal Residual Disease for Postoperative Recurrence and Adjuvant PD-1 Inhibitor in Hepatocellular Carcinoma: A Prospective, Multicenter Study
Brief Title: Predictive Value of Minimal Residual Disease for Postoperative Recurrence and Adjuvant PD-1 Inhibitor in HCC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, Wan-Guang Zhang, Professor, Tongji Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHALLENGE-04
Record Dates: First submitted 2025-12-24; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: HCC; Minimal Residual Disease; Recurrence
MeSH Terms: conditions — Neoplasm, Residual; Recurrence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative active monitoring cohort (Active Comparator): The postoperative active monitoring cohort collected a single blood sample for MRD monitoring before the surgery, and then dynamically collected blood samples for MRD monitoring at each follow-up visit after the surgery. This cohort only received active monitoring after the surgery.
  Interventions: Other: Active monitoring
- Postoperative PD-1 inhibitor adjuvant therapy cohort (Experimental): The postoperative PD-1 inhibitor-adjuvant cohort collected one blood sample for MRD monitoring before surgery, and dynamically collected blood samples for MRD monitoring at each follow-up visit after surgery. This cohort received only regular PD-1 inhibitor-assisted treatment after surgery.
  Interventions: Drug: Adjuvant PD-1 inhibitors

INTERVENTIONS:
Drug: Adjuvant PD-1 inhibitors — The patients in the postoperative adjuvant treatment cohort received regular PD-1 inhibitor adjuvant therapy (Sintilimab), once every 21 days, for a total of 8 times, and undergoing dynamic MRD testing.
  Arms: Postoperative PD-1 inhibitor adjuvant therapy cohort
Other: Active monitoring — The patients in the active monitoring cohort only received regular follow-up and MRD testing after the surgery.
  Arms: Postoperative active monitoring cohort

SUMMARY:
Hepatocellular carcinoma (HCC) is a leading global cause of cancer-related mortality. While curative resection is pivotal, high postoperative recurrence rates remain a major challenge. Adjuvant immune checkpoint inhibitors (ICIs) show promise in improving outcomes, but biomarkers to identify patients who will benefit are lacking. Current clinicopathological risk factors for minimal residual disease (MRD) are suboptimal in sensitivity and specificity.

Circulating tumor DNA (ctDNA) analysis, reflecting real-time tumor dynamics, offers a promising approach for MRD detection. This study focuses on the methylation status of GNB4 and Riplet-genes located within HCC-associated CpG islands-using a bespoke bisulfite-conversion and qPCR assay to sensitively detect methylated alleles, thereby enabling MRD monitoring.

To clinically validate this approach, we will conduct a prospective, multicenter cohort study assessing the predictive value of serial *GNB4/Riplet* methylation testing for recurrence and adjuvant therapy benefit.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is a leading global malignancy and a primary cause of mortality in patients with chronic liver disease. While curative resection offers a critical treatment strategy, postoperative recurrence remains a major obstacle. Emerging evidence suggests adjuvant therapy with immune checkpoint inhibitors (ICIs), such as PD-1/PD-L1 inhibitors, may improve disease-free survival; however, identifying the patient subgroup most likely to benefit remains challenging. Theoretically, patients at high risk for minimal residual disease (MRD) post-surgery represent the ideal target for adjuvant treatment. Current clinical practice relies on indirect pathological surrogates of MRD-such as microvascular invasion, poor differentiation, or satellite nodules-which lack sufficient sensitivity and specificity.

Cell-free DNA (cfDNA), with its short half-life, dynamically mirrors tumor evolution, making it a promising tool for monitoring recurrence. The genes GNB4 and Riplet are located within CpG islands strongly associated with hepatocarcinogenesis. We developed specific primers and fluorescent probes targeting their bisulfite-converted sequences to enable selective PCR-based detection of methylated alleles. Monitoring MRD via *GNB4/Riplet* methylation status thus offers a potential method for dynamic assessment of tumor progression and recurrence, optimizing patient risk stratification and guiding therapeutic decisions.

To evaluate this approach, we will conduct a prospective, multi-center cohort study to investigate the predictive value of MRD for recurrence and adjuvant therapy benefit. The study comprises two cohorts: 1) an Active Surveillance Cohort, undergoing a pre-operative MRD assessment followed by regular post-operative surveillance and serial MRD testing; and 2) an Adjuvant Therapy Cohort, receiving pre-operative MRD assessment followed by standard adjuvant PD-1 inhibitor therapy alongside serial MRD monitoring. This study aims to validate a more effective tool for predicting recurrence and to identify patients most likely to benefit from adjuvant immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 years, inclusive, regardless of gender.
* Newly diagnosed, treatment-naïve patients with HCC.
* Received radical treatments, such as liver resection or microwave ablation.
* Combine at least one of the risk factors for tumor recurrence, such as microvascular/macrovascular invasion, poor differentiation, satellite nodules, multiple tumors, and tumor diameter greater than 5 cm.
* Child-Pugh liver function score ≤ 7.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Absence of severe organic diseases affecting the heart, lungs, brain, or other major organs.

Exclusion Criteria:

* History of other malignancies.
* Recurrent HCC.
* Prior systemic therapy for HCC.
* Unable to complete the follow-up and dynamic MRD monitoring.
* Having an immune deficiency disorder.
* Allergic to PD-1 inhibitors or unable to tolerate related treatments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival(DFS) | From date of surgery until the date of first documented recurrence or date of death from any cause, whichever came first, assessed up to 60 months.
  DFS is defined as the time from surgery to the first recurrence. The difference in DFS between the two cohorts is compared.

SECONDARY OUTCOMES:
Overall survival(OS) | From date of surgery until the date of death from any cause, assessed up to 96 months.
  OS is defined as the time from surgery to the date of death.

OTHER OUTCOMES:
Association between dynamic Minimal Residual Disease (MRD) status and Disease-free survival (DFS) | From baseline up to 24 months.
  The predictive efficacy of dynamic MRD monitoring for recurrence. MRD will be assessed in peripheral blood samples at specified time points. The association between MRD status (positive/negative) and DFS will be quantified using Cox proportional hazards regression. The primary analysis will evaluate the hazard ratio for recurrence or death in MRD-positive vs. MRD-negative participants.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Hepato-Pancreato-Biliary Surgery, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China